CLINICAL TRIAL: NCT04097496
Title: Multi-Site Cluster, Randomized Proof of Concept Trial to Study the Effects of the ACT OUT! Social Issue Theater Program on Social-Emotional Competence and Bullying in Youth and Adolescents
Brief Title: Effects of ACT OUT! Social Issue Theater on Youth and Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic and related school policies.
Sponsor: Indiana University (Other)
Collaborators: Claude McNeal Productions (Unknown); Lilly Endowment, Inc. (Unknown)
Responsible Party: Principal Investigator, Jon Agley, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019 0543; 161999 (Other: Indiana University)
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Social Competence; Bullying
MeSH Terms: conditions — Social Skills; Bullying

STUDY DESIGN:
Intervention Model Description: The ACT OUT! Trial is designed as a proof-of-concept, cluster, randomized, superiority trial with two parallel groups. Randomization will be performed within clusters with a 1:1 allocation.
Who Masked: Outcomes Assessor
Masking Description: Because of the nature of the ACT OUT! trial, blinding of the trial participants, school officials, and members of Claude McNeal Productions is not possible. Further, since data management will occur via the primary research team, group identity cannot realistically be masked. However, we have included two statistical consultants - one internal to the university and one external to the university - who will be asked to verify all analyses using masked group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Act Out! Intervention (Experimental): Eligible classrooms will be randomized to attend a 1-hour ACT OUT! interactive, semi-improvisational psychodrama performance. The ACT OUT! intervention is an established theater program (https://www.claudemcnealproductions.com/act-out-ensemble/). The ACT OUT! production will include three to five vignettes paired with moderated discussions between the audience and the actors, the latter who will remain partly in character for the duration of the intervention. Vignettes will be different for each grade level included in the study (4th, 7th, and 10th). Public documentation of the guidelines for the ACT OUT! intervention will be made available as a supplemental file attached to the primary outcomes paper for the study.
  Interventions: Behavioral: Act Out! Intervention
- Control (No Intervention): Classrooms randomized to this arm will continue with their school day as normal, except that they will complete the data collection tools.

INTERVENTIONS:
Behavioral: Act Out! Intervention — Data included in the description of the intervention arm.
  Arms: Act Out! Intervention

SUMMARY:
The ACT OUT! Trial is designed as a proof-of-concept, cluster, randomized, superiority trial with two parallel groups. Although the unit of measurement is student, the unit of randomization is classroom, stratified by school. For each grade, an even number of classrooms will be selected from each school; half of the selected classrooms will be randomly assigned to intervention arm, whereas the other half will be assigned to control arm. This way, sociodemographic and school-level factors will be made approximately comparable between intervention and control arms.

DETAILED DESCRIPTION:
This study will be an assessment of the ACT OUT! Social Issue Theater program as a universal social and emotional learning (SEL) intervention targeting social-emotional competence (SEC) and bullying in elementary, middle, and high school students. ACT OUT! is an existing program that has been performed in various forms by professionally-trained members of an acting ensemble since 1995. The present iteration consists of three distinct scenarios per grade range (elementary, middle, and high) that present age-appropriate improvisational drama illustrating issues related to SEL and bullying, including facilitated discussion with the actors, who remain in character. The program lasts approximately one hour (scenario descriptions and a fidelity checklist for SEL/bullying elements will be made available as supplemental files).

SEL curricula typically consist of manualized and/or structured classroom or multicomponent programs taking place over time; the median number of sessions within an SEL program in a meta-analysis of 213 SEL studies was 24. At one hour in duration, ACT OUT! is substantially shorter and is performed by professional actors - meeting the goal of reduced school resource costs for SEL programming, but potentially raising concerns about whether such a dose could reasonably be expected to produce an effect. Underlying this study is a supposition that unique properties of a dramatic performance specifically may trigger SEL responses. In Aristotle's Poetics, which is the first known work on dramatic theory, it is written that a dramatic tragedy (in the Aristotelian sense) is designed to arouse certain feelings, "wherewith to accomplish catharsis of… emotions." This precise mechanism underlies the development of psychodrama as a psychotherapeutic intervention, as combined action and verbalization can present a situation "freed from the restricting stereotyped residues of past experience." Recent studies and meta-analyses have examined psychodrama as a means of prevention and/or behavior change with generally positive findings. Researchers have also found that youth report that they enjoy psychodramatic elements as part of a larger prevention curriculum. However, no studies have measured any outcomes of a psychodramatic SEL experience.

This will be the first study to examine whether a short dose of interactive psychodrama can affect SEC metrics and bullying experiences in schoolchildren. In responding to recent criticism of SEL studies, the investigators have chosen to utilize the SPIRIT 2013 clinical trial guidelines in developing this protocol to promote rigor, reproducibility, and transparency.

ELIGIBILITY:
Inclusion Criteria:

* Classrooms must be comprised of 4th grade (Elementary), 7th grade (Middle), or 10th grade (High) students

Exclusion Criteria:

* Participants and their parents or legal guardians will review study procedures. Parents or guardians may opt out on behalf of their dependents, and participants may themselves opt out.
* If a given grade within a school has an odd number of classrooms, one classroom randomly will be excluded from participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1537 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Social-Emotional Competence | Separately, 2 weeks post-intervention, and 3 months post-intervention
  Computed from the Delaware Social Emotional Competency Scale (DSECS-S). The score is averaged from Likert-type data (e.g., one overall score will be computed from 12 questions). The score ranges from '1' to '4' - some items will be reverse coded, so that a '4' is consistently the optimal score across questions and for the total scale value.
Change from Baseline Bullying Prevalence (self-report) | Separately, 2 weeks post-intervention, and 3 months post-intervention
  Bullying activity (being bullied and bullying) via two parallel 13-item scales on the Bullying and Cyberbullying Scale for Adolescents (BCS-A). This scale captures frequency data and so is interpretable on its face (e.g., # instances of a behavior or observation).
Change from Baseline Bullying Prevalence (objective) | 3 months post-intervention
  Disciplinary referrals for bullying (aggregated, not individual)

SECONDARY OUTCOMES:
Change from Baseline Social-Emotional Competence Sub-Domains (7th and 10th grades only) | Separately, 2 weeks post-intervention, and 3 months post-intervention
  Social awareness, emotion regulation, relationship skills, and responsible decision-making as measured via 4 sub-scales of the Washoe County School District Social-Emotional Competency Assessment. For each sub-scale, the score is averaged from Likert-type data (e.g., one overall score will be computed from 3-5 questions). The score ranges from '1' to '4' - a '4' is consistently the optimal score across questions and for the total scale value.
Receptivity to the Act Out! Intervention | 2 weeks post-intervention
  Subjective receptivity to the intervention (e.g., enjoyment) as measured by response items from Dent et al. (1998). This scale *does not* have a specific name. It measures the following characteristics of receptivity to the intervention: whether it was enjoyable, interesting, a waste of time, boring, understandable, difficult to understand, believable, important, and helpful. Each item is measured using a Likert-type scale. The score ranges from '1' to '4' - some items will be reverse coded, so that a '4' is consistently the optimal score across questions and for the total scale value.
Frequency of Truancy/Absenteeism | 3 months post-intervention
  Data for clusters from district records (aggregated, not individual). These data already exist. No individual-level data will be utilized, only aggregated frequency of truancy/absenteeism.
Academic Performance using standard Grade Point Average | 3 months post-intervention
  Data for clusters from district records (aggregated, not individual); grade point average normalized to a 4.0 grading scale (where 4.0 is an A and 1.0 is an F).

CONTACTS AND LOCATIONS:
Locations (1):
- Claude McNeal Productions, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in study publications will be made available in fully de-identified form. The study protocol will be published in an open-access journal and will include the statistical analysis plan, per SPIRIT 2013 recommendations.
  All forms related to recruitment and protocol execution will also be made available as supplemental files in appropriate outcome publications. The analytic code for each outcome publication will be published as a supplemental file with the corresponding paper.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available at the time of publication.
Access Criteria: Data will be open-access.

REFERENCES:
- [Background] Claude McNeal Productions. Act Out Ensemble [Internet]. Claude McNeal Productions. 2019 [cited 11 September 2019]. Available from: https://www.claudemcnealproductions.com/act-out-ensemble/
- [Background] Durlak JA, Weissberg RP, Dymnicki AB, Taylor RD, Schellinger KB. The impact of enhancing students' social and emotional learning: a meta-analysis of school-based universal interventions. Child Dev. 2011 Jan-Feb;82(1):405-32. doi: 10.1111/j.1467-8624.2010.01564.x. PMID 21291449
- [Background] Rosenstein L. On Aristotle and thought in drama. Critical Inquiry. 1977;3(3):543-65.
- [Background] Davies MH. The origins and practice of psychodrama. Br J Psychiatry. 1976 Sep;129:201-6. doi: 10.1192/bjp.129.3.201. PMID 786420
- [Background] Krahé B, Knappert L. A group-randomized evaluation of a theatre-based sexual abuse prevention programme for primary school children in Germany. J Community Appl Soc Psychol. 2009;19(4):321-9.
- [Background] Lauby JL, LaPollo AB, Herbst JH, Painter TM, Batson H, Pierre A, Milnamow M. Preventing AIDS through live movement and sound: Efficacy of a theater-based HIV prevention intervention delivered to high-risk male adolescents in juvenile justice settings. AIDS Educ Prev. 2010 Oct;22(5):402-16. doi: 10.1521/aeap.2010.22.5.402. PMID 20973661
- [Background] Lightfoot AF, Taboada A, Taggart T, Tran T, Burtaine A. 'I learned to be okay with talking about sex and safety': assessing the efficacy of a theatre-based HIV prevention approach for adolescents in North Carolina. Sex Educ. 2015;15(4):348-363. doi: 10.1080/14681811.2015.1025947. PMID 26300693
- [Background] Joronen K, Konu A, Rankin HS, Astedt-Kurki P. An evaluation of a drama program to enhance social relationships and anti-bullying at elementary school: a controlled study. Health Promot Int. 2012 Mar;27(1):5-14. doi: 10.1093/heapro/dar012. Epub 2011 Mar 7. PMID 21385761
- [Background] Cheadle A, Cahill C, Schwartz PM, Edmiston J, Johnson S, Davis L, Robbins C. Engaging youth in learning about healthful eating and active living: an evaluation of Educational Theater Programs. J Nutr Educ Behav. 2012 Mar-Apr;44(2):160-5. doi: 10.1016/j.jneb.2011.06.005. Epub 2011 Nov 25. PMID 22118997
- [Background] Belknap RA, Haglund K, Felzer H, Pruszynski J, Schneider J. A theater intervention to prevent teen dating violence for Mexican-American middle school students. J Adolesc Health. 2013 Jul;53(1):62-7. doi: 10.1016/j.jadohealth.2013.02.006. Epub 2013 Apr 11. PMID 23583507
- [Background] Joronen K, Rankin SH, Astedt-Kurki P. School-based drama interventions in health promotion for children and adolescents: systematic review. J Adv Nurs. 2008 Jul;63(2):116-31. doi: 10.1111/j.1365-2648.2008.04634.x. PMID 18537845
- [Background] Sussman SY. Evaluating the efficacy of Project TND: Evidence from seven research trials. In: Scheier LM, editor. Handbook of adolescent drug use prevention: Research, intervention strategies, and practice. Washington DC: American Psychological Association; 2015. p. 159-76.
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Mantz LS, Bear GC, Yang C, Harris, A. The Delaware Social-Emotional Competency Scale (DSECS-S): Evidence of validity and reliability. Child Indic Res. 2018;11(1):137-57.
- [Background] Thomas HJ, Scott JG, Coates JM, Connor JP. Development and validation of the Bullying and Cyberbullying Scale for Adolescents: A multi-dimensional measurement model. Br J Educ Psychol. 2019 Mar;89(1):75-94. doi: 10.1111/bjep.12223. Epub 2018 May 3. PMID 29726005
- [Background] Dent CW, Sussman S, Hennesy M, Galaif ER, Stacy AW, Moss M, Craig S. Implementation and process evaluation of a school-based drug abuse prevention program: Project Towards No Drug Abuse. J Drug Educ. 1998;28(4):361-75. doi: 10.2190/UFY9-WHXX-AFC1-RXB1. PMID 10097485
- [Derived] Agley J, Jun M, Eldridge L, Agley DL, Xiao Y, Sussman S, Golzarri-Arroyo L, Dickinson SL, Jayawardene W, Gassman R. Effects of ACT Out! Social Issue Theater on Social-Emotional Competence and Bullying in Youth and Adolescents: Cluster Randomized Controlled Trial. JMIR Ment Health. 2021 Jan 6;8(1):e25860. doi: 10.2196/25860. PMID 33338986
- [Derived] Agley J, Jayawardene W, Jun M, Agley DL, Gassman R, Sussman S, Xiao Y, Dickinson SL. Effects of the ACT OUT! Social Issue Theater Program on Social-Emotional Competence and Bullying in Youth and Adolescents: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2020 Apr 13;9(4):e17900. doi: 10.2196/17900. PMID 32281541